CLINICAL TRIAL: NCT05102344
Title: Animal Assisted Intervention With Dogs for Children With Attention Deficit/Hyperactivity Disorder; Exploring Candidate Physiological Markers of Response to AAI
Brief Title: Animal Assisted Intervention With Dogs for Children With ADHD
Acronym: PACK-PM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sabrina E. Brierley Schuck, Ph.D., Associate Professor in Residence, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20206069; R21HD103422 (NIH)
Record Dates: First submitted 2021-10-08; First posted 2021-11-01 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Animal Assisted Intervention; Social Skills Training
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Lab assistants responsible for processing biological samples of interest and the principal statistician are blind to identifying participant information and group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychosocial Treatment as Usual (Active Comparator): Participants assigned to the active comparator arm will receive active non-pharmacological treatment utilizing behavioral social skills training strategies previously found to be effective in reducing symptoms of ADHD and improving social skills for children with ADHD
  Interventions: Behavioral: Behavioral Social Skills Training
- Animal Assisted Intervention (Experimental): Participants assigned to the experimental arm will receive active non-pharmacological treatment utilizing behavioral social skills training strategies previously found to be effective in reducing symptoms of ADHD and improving social skills for children with ADHD accompanied by live therapy dogs
  Interventions: Behavioral: Animal Assisted Intervention

INTERVENTIONS:
Behavioral: Behavioral Social Skills Training — Behavioral Social Skills Training treatment as usual will include small group semi-structured play, didactic instruction and role-play of basic social skills, including assertion, ignoring provocation, accepting consequences, problem solving, following directions, and self-regulation.
  Arms: Psychosocial Treatment as Usual
Behavioral: Animal Assisted Intervention — Behavioral Social Skills Training treatment as usual will include small group semi-structured play, didactic instruction and role-play of basic social skills, including assertion, ignoring provocation, accepting consequences, problem solving, following directions, and self-regulation accompanied by trained therapy dogs
  Arms: Animal Assisted Intervention

SUMMARY:
This pilot study aims to replicate results of a previously studied novel, non-pharmacological psychosocial intervention for children with ADHD, utilizing an Animal Assisted Intervention with therapy dogs combined with traditional social skills training (AAI) compared to psychosocial treatment as usual with social skills training alone (TAU). This study also aims to determine if candidate physiological markers of HPA axis and ANS activity differ between groups and if these markers moderate response to the interventions.

DETAILED DESCRIPTION:
Attention-Deficit/Hyperactivity Disorder (ADHD) is the most commonly occurring neurodevelopmental disorder in the United States, with current prevalence rates between 8% and 11%, up from an estimated 5% in 2003. Despite decades of research, individuals with ADHD continue to be at significantly greater risk for poor life outcomes compared to non-affect peers. Evidence-based interventions for ADHD include stimulant medications and psychosocial treatments, but these practices are not always feasible or acceptable due to adverse side-effects, cost, availability, and poor treatment adherence. ADHD is considered to be a result of a physiological disruption of select catecholaminergic systems (e.g. dopamine and norepinephrine) and related under-arousal of cognitive functions of the pre-frontal cortex involved in executive functioning (EF). Research indicates that AAI with dogs is effective for improving social-behavioral outcomes related to EF deficits. The mechanisms by which AAI improves outcomes for this group and mediators of these outcomes, however, is not yet understood. These gaps in understanding hinder progress in the application of AAI, limiting the acceptability and availability of this integrative health care practice. Recent research in other populations suggests that AAI acts on hypothalamic-pituitary-adrenal (HPA) axis activity, reducing physiological stress Children with ADHD, however, present with different Autonomic Nervous System (ANS) response patterns when compared to typically developing children and children with other mental health disorders and this phenomenon points to altered physiological activity in response to stress, social feedback, and emotional stimuli when compared to their peers. The bio-social mechanistic hypothesis proposed in this study contends that dogs may elicit physiological responses related to cognitive arousal of EF systems, thereby enhancing response to treatment in children with ADHD. Furthermore, given the heterogeneity of impairment and high comorbidity with other mental health disorders among children with ADHD and the prevalence of ADHD across cultures, race and ethnicity, individual differences in response to AAI and in child/animal interaction may potentially mediate response to AAI. This research will explore these gaps by: 1) replicating findings from a previous AAI Randomized Controlled Trial on social-behavioral outcomes, 2) exploring candidate physiological responses to AAI over time, and 3) ascertaining if individual differences during AAI mediate primary and/or exploratory main outcomes. This study hypothesizes AAI will result in enhanced social-behavioral outcomes and improved diurnal patterns of HPA and ANS for these children. Furthermore, it is suspected acute physiological responses to AAI (markers of HPA & ANS) and social interaction quality (child/child and child/dog) will mediate main outcomes. To explore these hypotheses, the investigators will conduct an exploratory parallel-group randomized controlled clinical trial with 48 young children with ADHD, participating in psychosocial intervention with or without AAI using a previously manualized AAI model developed and found successful in prior work. This work will yield the first information on candidate mechanisms thought to play an important role in AAI for children with ADHD, thus laying foundations for later submission of a fully powered, multi-site randomized clinical trial aimed to better inform approaches refined for this group, and promote acceptability and generalizability of AAI with children with special needs.

ELIGIBILITY:
Inclusion Criteria:

* Meets research criteria for a diagnosis of ADHD based on the Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS)
* Has never taken stimulant medication or has had at least a 6 week 'wash-out' period from stimulant medicines not related to enrollment in the study.

Exclusion Criteria:

* Is currently taking stimulant medications or has taken stimulant medications within the last 6 weeks
* Allergy to dogs
* Significant fear of dogs
* Family history or history of cruelty to animals
* Meets research criteria for a diagnosis of Autism Spectrum Disorder (ASD) based on the K-SADS and Autism Specturm Rating Scale (ASRS) total raw score in the 'severe range'
* Meets research criteria for a diagnosis of Major Depressive Disorder on the K-SADS
* Meets research criteria for a diagnosis of Schizophrenia on the K-SADS

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina EB Schuck, Ph.D., Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schuck SEB, Zeiler CN, Stehli A, Steinhoff LA, Stokes RY, Jeffrey SE, Granger DA. Acute salivary cortisol response in children with ADHD during psychosocial intervention with and without therapy dogs. Front Psychiatry. 2024 Oct 24;15:1476522. doi: 10.3389/fpsyt.2024.1476522. eCollection 2024. PMID 39512897

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Psychosocial Treatment as Usual | Animal Assisted Intervention
Started | 19 | 20
Completed | 19 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Psychosocial Treatment as Usual | Animal Assisted Intervention | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 20 | 39
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 8.409 [7 to 9] | 8.207 [7 to 9] | 8.305 [7 to 9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 15 | 16 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 16 | 13 | 29
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 14 | 28
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 39
Attention Deficit Hyperactivity Disorder-Rating Scale [Mean (Standard Deviation); unit: units on a scale] — The Attention Deficit/Hyperactivity Disorder Rating Scale (ADHD-RS-5; DuPaul) measures parent ratings of severity of ADHD symptoms using a 4-point Likert Scale, rating 18 items with ratings from 0-3. The total score reported represents the total for the 18 itmes, with a range of 0 to 54, with higher scores indicating greater impairment from symptoms. Population: Implementation error. Scale was not captured at two baseline visits.
  units on a scale
    number analyzed (Participants) | 19 | 18 | 37
    (all) | 41.84 (8.1) | 42.06 (7.9) | 41.9 (8.2)
Autism Spectrum Rating System (ASRS) [Mean (Standard Deviation); unit: units on a scale] — The Autism Spectrum Rating System, Short Form, Adapted 6-18 years (ASRS; Goldstein) is rating scale completed by parents utilizing a 5-point Likert scale (0-4) for 15 items measuring Autism symptom severity. Total values are converted to T-scores ranging from 28 to 85, with higher scores indicating greater symptoms severity, Population: Implementation error. Scale was not completed by three parents.
  units on a scale
    number analyzed (Participants) | 19 | 17 | 36
    (all) | 57.37 (9.1) | 56.82 (9.7) | 57.11 (9.6)
Wechsler Abbreviated Scale of Intelligence (WASI) [Mean (Standard Deviation); unit: units on a scale] — The Wechsler Abbreviated Scale of Intelligence, second edition (WASI-2;Wechsler) is a brief measure of general intelligence, or IQ test designed to assess specific and overall cognitive capabilities and is individually administered to children, adolescents and adults (ages 6-89), composed of 4 sub-scales with scores combined and transformed to an age standardized The test is based on a mean score of 100 and a standard deviation of 15, with scores typically ranging from 40 to 160, with greater scores representing higher or more proficient cognitive capabilities.
  units on a scale | 102.32 (10.3) | 105.65 (13.0) | 104.03 (12.7)
Test of Word Reading Efficiency (TOWRE) [Mean (Standard Deviation); unit: units on a scale] — The Test of Word Reading Efficiency, second edition (TOWRE-2;Torgesen, Wagner and Rashotte) is measure of reading skills for children ages 6-24, composed of 167 questions across two scales. Sub-scale scores are combined for a total score and transformed to age-based standardized scores. The test is based on a mean score of 100 and a standard deviation of 15, with total scores of less than 70 considered to be 'very poor' and scores and scores over 130 as 'very superior' with average scores falling between 90-110. Population: One participant was unable to complete the assessment.
  units on a scale
    number analyzed (Participants) | 19 | 19 | 38
    (all) | 97.63 (13.8) | 92.8 (15.9) | 95.24 (15.8)
Social Responsiveness Scale (SRS-2) [Mean (Standard Deviation); unit: T-Score] — The Social Responsiveness Scale, second edition, (SRS-2: Constantino) measures parent ratings of symptoms of Autism Spectrum Disorder for individuals (preschool to adulthood). It is a 65-item, 4-point Likert rating scale with item scores ranging (1-4). Total scores are summed from 5 sub-scales and transformed to a Total T-score reported above. The population mean for the Total T-score value is 50 with a standard deviation of 10, with scores of 59 and below considered normal, and higher scores indicating a greater likelihood of a clinical diagnosis of ASD. Population: This measure was not gathered for first three participants and one additional parent refused.
  T-Score
    number analyzed (Participants) | 18 | 17 | 35
    (all) | 62.06 (10.95) | 61.53 (10.9) | 61.8 (10.77)
National Institutes of Health Toolkit-Flanker Task [Mean (Standard Deviation); unit: units on a scale] — The National Institutes of Health Toolkit, Flanker Inhibitory Control and Attention Test measures inhibitory control and attention. Scores are based on both accuracy and reaction time, and the final score is determined by an algorithm that considers both. If accuracy is less than or equal to 80%, the score is based on accuracy alone. For those with accuracy greater than 80%, the score combines accuracy and reaction time. The age-adjusted scale scores have a mean of 100 and a standard deviation of 15, with higher scores representing more inhibitory control and better attention. Population: One participant refused to complete the assessment task.
  units on a scale
    number analyzed (Participants) | 19 | 19 | 38
    (all) | 90.79 (10.7) | 88.68 (12.5) | 89.74 (11.6)
NIH Toolkit List Sort Task [Mean (Standard Deviation); unit: units on a scale] — The National Institutes of Health Toolkit, List Sorting Working Memory Test measures working memory skills or ability to hold and manipulate information. The age-adjusted scale scores have a mean of 100 and a standard deviation of 15, with higher scores representing better working memory performance. Population: Two participants refused, were absent, or unable to complete the assessment.
  units on a scale
    number analyzed (Participants) | 19 | 18 | 37
    (all) | 90.58 (16.0) | 96.89 (14.9) | 93.7 (15.2)
NIH Toolkit Dimensional Change [Mean (Standard Deviation); unit: units on a scale] — The National Institutes of Health Toolkit, Dimensional Change Card Sort test measures cognitive flexibility and attention. The age-adjusted scale scores have a mean of 100 and a standard deviation of 15, with higher scores representing better cognitive flexibility. Population: One participants refused, were absent, or unable to complete the assessment.
  units on a scale
    number analyzed (Participants) | 19 | 19 | 38
    (all) | 91.74 (12.1) | 92.21 (12.5) | 91.97 (12.3)
Social Skills Improvement System-Social Skills Scub-scale [Mean (Standard Deviation); unit: units on a scale] — The Social Skills Improvement System Rating Scales, parent version, social skills sub-scale (SSIS-RS; Gresham) is a norm-referenced rating form used to assess social skills in children and adolescents aged 3-18. The Social Skills sub-scale is composed of 46-items and utilizes a 4-point Likert scale, with item scores ranging from 0-3. The total sub-scale summed score is age-adjusted and scaled scores have a mean of 100 and a standard deviation of 15, with higher scores representing better social skills. Population: Parent rater neglected to complete rating scales for 4 participants
  units on a scale
    number analyzed (Participants) | 18 | 17 | 35
    (all) | 85.79 (13.9) | 83.95 (9.1) | 84.85 (11.85)
Social Skills Improvement System-Problem Behaviors [Mean (Standard Deviation); unit: units on a scale] — The Social Skills Improvement System Rating Scales, parent version, problem behaviors sub-scale (SSIS-RS; Gresham) is a norm-referenced rating form used to assess problem behaviors in children and adolescents aged 3-18. The Problem Behaviors sub-scale is composed of 33-items and utilizes a 4-point Likert scale, with item scores ranging from 0-3. The total sub-scale summed score is age-adjusted and scaled scores have a mean of 100 and a standard deviation of 15, with higher scores representing more problematic behavior. Population: parent neglected to complete rating scale for 4 participants
  units on a scale
    number analyzed (Participants) | 18 | 17 | 35
    (all) | 122.58 (15.56) | 122.40 (13.89) | 122.49 (14.53)
Self-Perception Profile for Children (Harter) [Mean (Standard Deviation); unit: units on a scale] — The Self-Perception Profile for Children (SPPC; Harter) uses a 4-point Likert scale, where each item is scored from 1 to 4. The SPPC measures self-perceptions across six domains: Scholastic Competence, Social Acceptance, Athletic Competence, Physical Appearance, Behavioral Conduct, and Global Self-Worth, with a total score summing and averaging 36 items with a total score of 1 being the lowest perceived competence or adequacy, and a score of 4 represents the highest level of competence or adequacy.
  units on a scale | 3.05 (0.601) | 3.08 (0.514) | 3.06 (0.605)
Diurnal Salivary Cortisol Levels at Baseline [Mean (Standard Deviation); unit: ug/mL per day] — Cortisol is a stress-sensitive hormone which follows a diurnal cycle. Diurnal change in cortisol is typically measured as a negative slope value with average scores often around -1.00, with steeper (more negative) scores associated with well-being and flatter diurnal cortisol slopes associated with chronic psychosocial stress and poor outcomes in past theory and research. Secreted cortisol levels were measured from saliva samples were collected at three time points (awakening, morning, bedtime) across two days before intervention to calculate baseline group mean slope. Population: One participant refused to provide a saliva sample at this time point.
  ug/mL per day
    number analyzed (Participants) | 18 | 20 | 38
    (all) | -.13959 (.06) | -.14196 (.07) | -.1408 (.06)
Diurnal Salivary Alpha-Amylase at Baseline [Mean (Standard Deviation); unit: u/mL per day] — Salivary Alpha Amylase (sAA) is an enzyme marker of the autonomic/sympathetic nervous system (ANS/SNS) steadily rises over the day. Diurnal change is measured as a positive slope value. Steeper slope indicates faster increase in sAA levels and has been associated with poor health outcomes. Secreted sAA levels were measured from saliva collected at three time points (awakening, morning, bedtime) over two days before intervention to calculate baseline group mean slope. Interpretation of values requires consideration of the context and was collected at baseline for comparison to other variables. Population: One participant refused to provide a saliva sample at this collection point.
  u/mL per day
    number analyzed (Participants) | 18 | 20 | 38
    (all) | 4.90406 (14.95) | 8.1836 (14.83) | 6.63 (14.9)
Salivary Uric Acid at Baseline [Mean (Standard Deviation); unit: mg/dL] — Salivary Uric Acid (sUA) is a biomarker that may be associated with increases in blood pressure in response to stress and self-perception of power suggesting that sUA may play an important role in self-competence. Baseline concentration of sUA was measured from saliva collected at one time time point prior to intervention. Interpretation of values requires consideration of the context and was collected at baseline for comparison to other variables. Population: One participant refused to provide a saliva sample at this collection point.
  mg/dL
    number analyzed (Participants) | 18 | 20 | 38
    (all) | 3.51 (2.51) | 3.34 (2.29) | 3.44 (2.40)

OUTCOME MEASURES:

1. Primary Outcome: ADHD-Rating Scale (ADHD-RS) at 8 Weeks
Description: Attention Deficit/Hyperactivity Rating Scale for Parents is a categorical and dimensional parent and teacher ratings of symptoms of inattention, hyperactivity, and impulsivity (min: 0.00, max: 54.00; lower scores indicate less impairment).
Time Frame: At 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychosocial Treatment as Usual | Animal Assisted Intervention
Number analyzed (Participants) | 19 | 20
units on a scale | 29.0 (9.1) | 23.9 (8.44)

2. Primary Outcome: ADHD-Rating Scale (ADHD-RS) at 16 Weeks Follow-up
Description: as for outcome 1
Time Frame: At 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychosocial Treatment as Usual | Animal Assisted Intervention
Number analyzed (Participants) | 17 | 19
units on a scale | 28.29 (12.0) | 24.26 (7.93)

3. Primary Outcome: Self-Perception Profile for Children (SPPC) at 8 Weeks
Description: The Self-Perception Profile for Children (SPPC; Harter) uses a 4-point Likert scale, where each item is scored from 1 to 4. The SPPC measures self-perceptions across six domains: Scholastic Competence, Social Acceptance, Athletic Competence, Physical Appearance, Behavioral Conduct, and Global Self-Worth, with a total score summing and averaging 36 items with a total score of 1 being the lowest perceived competence or adequacy, and a score of 4 represents the highest level of competence or adequacy.
Time Frame: At 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychosocial Treatment as Usual | Animal Assisted Intervention
Number analyzed (Participants) | 18 | 20
units on a scale | 2.981 (.613) | 3.142 (.463)

4. Primary Outcome: Self-Perception Profile for Children (SPPC) at 16 Weeks
Description: as for outcome 3
Time Frame: At 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychosocial Treatment as Usual | Animal Assisted Intervention
Number analyzed (Participants) | 19 | 19
units on a scale | 2.956 (0.673) | 3.236 (0.301)

5. Primary Outcome: Social Responsiveness Scale (SRS-2) at 8 Weeks
Description: The Social Responsiveness Scale, second edition, (SRS-2: Constantino) measures parent ratings of symptoms of Autism Spectrum Disorder for individuals (preschool to adulthood). It is a 65-item, 4-point Likert rating scale with item scores ranging (1-4). Total scores are summed from 5 sub-scales and transformed to a Total T-score reported above. The population mean for the Total T-score value is 50 with a standard deviation of 10, with scores of 59 and below considered normal, and higher scores indicating a greater likelihood of a clinical diagnosis of ASD.
Time Frame: At 8 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Psychosocial Treatment as Usual | Animal Assisted Intervention
Number analyzed (Participants) | 18 | 17
T-score | 57.89 (9.5) | 60.80 (11.31)

6. Primary Outcome: Social Responsiveness Scale (SRS-2) at 16 Weeks
Description: as for outcome 5
Time Frame: At 16 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Psychosocial Treatment as Usual | Animal Assisted Intervention
Number analyzed (Participants) | 18 | 17
T-score | 57.16 (12.00) | 58.90 (9.97)

7. Primary Outcome: Social Skills Improvement System Rating Scales (SSIS-RS) Social Skills at 8 Weeks
Description: The Social Skills Improvement System Rating Scales, parent version, social skills sub-scale (SSIS-RS; Gresham) is a norm-referenced rating form used to assess social skills in children and adolescents aged 3-18. The Social Skills sub-scale is composed of 46-items and utilizes a 4-point Likert scale, with item scores ranging from 0-3. The total sub-scale summed score is age-adjusted and scaled scores have a mean of 100 and a standard deviation of 15, with higher scores representing better social skills.
Time Frame: At 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychosocial Treatment as Usual | Animal Assisted Intervention
Number analyzed (Participants) | 19 | 20
units on a scale | 90.16 (14.50) | 87.80 (13.51)

8. Primary Outcome: Social Skills Improvement System Rating Scales (SSIS-RS) Social Skills at 16 Weeks
Description: as for outcome 7
Time Frame: At 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychosocial Treatment as Usual | Animal Assisted Intervention
Number analyzed (Participants) | 19 | 20
units on a scale | 89.84 (14.50) | 90.10 (12.64)

9. Primary Outcome: Social Skills Improvement System Rating Scale (SSIS-RS) Problem Behaviors at 8 Weeks
Description: The Social Skills Improvement System Rating Scales, parent version, problem behaviors sub-scale (SSIS-RS; Gresham) is a norm-referenced rating form used to assess problem behaviors in children and adolescents aged 3-18. The Problem Behaviors sub-scale is composed of 33-items and utilizes a 4-point Likert scale, with item scores ranging from 0-3. The total sub-scale summed score is age-adjusted and scaled scores have a mean of 100 and a standard deviation of 15, with higher scores representing more problematic behavior.
Time Frame: At 8 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychosocial Treatment as Usual | Animal Assisted Intervention
Number analyzed (Participants) | 19 | 20
units on a scale | 119.53 (15.85) | 117.55 (16.72)

10. Primary Outcome: Social Skills Improvement System Rating Scale (SSIS-RS) Problem Behaviors at 16 Weeks
Description: as for outcome 9
Time Frame: At 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychosocial Treatment as Usual | Animal Assisted Intervention
Number analyzed (Participants) | 19 | 20
units on a scale | 117.63 (17.41) | 114.10 (12.74)

11. Secondary Outcome: Diurnal Salivary Cortisol Levels at 8 Weeks
Description: Cortisol is a stress-sensitive hormone which follows a diurnal cycle. Diurnal change in cortisol is typically measured as a negative slope value with average scores often around -1.00, with steeper (more negative) scores associated with well-being and flatter diurnal cortisol slopes associated with chronic psychosocial stress and poor outcomes in past theory and research. Secreted cortisol levels were measured from saliva samples were collected at three time points (awakening, morning, bedtime) across two days at the end of the intervention (at 8 weeks from baseline) to calculate end of treatment group mean slopes.
Time Frame: At 8 weeks
Measure: Mean (Standard Deviation); unit: ug/mL per day
Arm/Group | Psychosocial Treatment as Usual | Animal Assisted Intervention
Number analyzed (Participants) | 18 | 20
ug/mL per day | -.1378 (0.08) | -.104 (.10)

12. Secondary Outcome: Diurnal Salivary Cortisol Levels at 16 Weeks
Description: Cortisol is a stress-sensitive hormone which follows a diurnal cycle. Diurnal change in cortisol is typically measured as a negative slope value with average scores often around -1.00, with steeper (more negative) scores associated with well-being and flatter diurnal cortisol slopes associated with chronic psychosocial stress and poor outcomes in past theory and research. Secreted cortisol levels were measured from saliva samples were collected at three time points (awakening, morning, bedtime) across two days at 8 weeks following end of the intervention (at 16 weeks from baseline) to calculate follow-up group mean slopes.
Time Frame: At 16 weeks
Measure: Mean (Standard Deviation); unit: ug/mL per day
Arm/Group | Psychosocial Treatment as Usual | Animal Assisted Intervention
Number analyzed (Participants) | 18 | 19
ug/mL per day | -.125 (.13) | -.136 (.10)

13. Secondary Outcome: Acute Salivary Cortisol Level (In-session Week 1)
Description: Cortisol is a stress-sensitive hormone which may be acutely sensitive to intervention. Secreted cortisol levels were measured from saliva samples collected at three time points during intervention sessions (arrival, 20 minutes later, and 40 minutes into the session) and to determine a mean cortisol level for each participant and calculate acute group mean averages at week 1.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Psychosocial Treatment as Usual | Animal Assisted Intervention
Number analyzed (Participants) | 19 | 20
ug/mL | .138 (.13) | .141 (.16)

14. Secondary Outcome: Acute Salivary Cortisol Level (In-session Week 4)
Description: Cortisol is a stress-sensitive hormone which may be acutely sensitive to intervention. Secreted cortisol levels were measured from saliva samples collected at three time points during intervention sessions (arrival, 20 minutes later, and 40 minutes into the session) and to determine a mean cortisol level for each participant and calculate acute group mean averages at week 4.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Psychosocial Treatment as Usual | Animal Assisted Intervention
Number analyzed (Participants) | 19 | 20
ug/mL | .103 (.051) | .102 (.059)

15. Secondary Outcome: Acute Salivary Cortisol Level (In-session Week 8)
Description: Cortisol is a stress-sensitive hormone which may be acutely sensitive to intervention. Secreted cortisol levels were measured from saliva samples collected at three time points during intervention sessions (arrival, 20 minutes later, and 40 minutes into the session) and to determine a mean cortisol level for each participant and calculate acute group mean averages at week 8.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Psychosocial Treatment as Usual | Animal Assisted Intervention
Number analyzed (Participants) | 18 | 18
ug/mL | .101 (.053) | .101 (.058)

16. Secondary Outcome: Alpha-Amylase From Saliva at 8 Weeks
Description: Salivary Alpha Amylase (sAA) is an enzyme marker of the autonomic/sympathetic nervous system (ANS/SNS) steadily rises over the day. Diurnal change is measured as a positive slope value. Steeper slope indicates faster increase in sAA levels and has been associated with poor health outcomes. Secreted sAA levels were measured from saliva collected at three time points (awakening, morning, bedtime) over two days before the last intervention intervention session (week 8) to calculate baseline group mean slope. Interpretation of values requires consideration of the context and was collected at 8-weeks for comparison to other variables.
Time Frame: At 8 weeks
Measure: Mean (Standard Deviation); unit: u/mL per day
Arm/Group | Psychosocial Treatment as Usual | Animal Assisted Intervention
Number analyzed (Participants) | 18 | 20
u/mL per day | 11.21 (17.6) | 17.21 (22.2)

17. Secondary Outcome: Alpha-Amylase From Saliva at 16 Weeks
Description: Salivary Alpha Amylase (sAA) is an enzyme marker of the autonomic/sympathetic nervous system (ANS/SNS) steadily rises over the day. Diurnal change is measured as a positive slope value. Steeper slope indicates faster increase in sAA levels and has been associated with poor health outcomes. Secreted sAA levels were measured from saliva collected at three time points (awakening, morning, bedtime) over two days before the follow-up session (week 16, or 8 weeks post-intervention) to calculate baseline group mean slope. Interpretation of values requires consideration of the context and was collected at 16-weeks for comparison to other variables.
Time Frame: At 16 weeks
Measure: Mean (Standard Error); unit: u/mL per day
Arm/Group | Psychosocial Treatment as Usual | Animal Assisted Intervention
Number analyzed (Participants) | 18 | 19
u/mL per day | 5.74 (16.7) | 13.37 (19.86)

18. Secondary Outcome: Acute Salivary Alpha-Amylase Level (In-session Week 1)
Description: Salivary alpha-amylase (sAA) is a biomarker of the autonomic/sympathetic nervous system (ANS/SNS) which may be acutely sensitive to intervention. Secreted sAA levels were measured from saliva samples collected at three time points during intervention sessions (arrival, 20 minutes later, and 40 minutes into the session) to determine a mean sAA level for each participant and calculate acute group mean averages at week 1.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: u/mL
Arm/Group | Psychosocial Treatment as Usual | Animal Assisted Intervention
Number analyzed (Participants) | 19 | 20
u/mL | 88.45 (46.4) | 88.93 (61.2)

19. Secondary Outcome: Acute Salivary Alpha-Amylase Level (In-session Week 4)
Description: Salivary alpha-amylase (sAA) is a biomarker of the autonomic/sympathetic nervous system (ANS/SNS) which may be acutely sensitive to intervention. Secreted sAA levels were measured from saliva samples collected at three time points during intervention sessions (arrival, 20 minutes later, and 40 minutes into the session) to determine a mean sAA level for each participant and calculate acute group mean averages at week 4.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: u/mL
Arm/Group | Psychosocial Treatment as Usual | Animal Assisted Intervention
Number analyzed (Participants) | 19 | 20
u/mL | 77.27 (51.4) | 84.68 (54.9)

20. Secondary Outcome: Acute Salivary Alpha-Amylase Level (In-session Week 8)
Description: Salivary alpha-amylase (sAA) is a biomarker of the autonomic/sympathetic nervous system (ANS/SNS) which may be acutely sensitive to intervention. Secreted sAA levels were measured from saliva samples collected at three time points during intervention sessions (arrival, 20 minutes later, and 40 minutes into the session) to determine a mean sAA level for each participant and calculate acute group mean averages at week 8.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: u/mL
Arm/Group | Psychosocial Treatment as Usual | Animal Assisted Intervention
Number analyzed (Participants) | 18 | 18
u/mL | 78.23 (61.5) | 94.34 (65.5)

21. Secondary Outcome: Acute Salivary Uric Acid Level (In-session Week 1)
Description: Salivary Uric Acid (sUA) is a biomarker that may be associated with increases in blood pressure in response to stress and self-perception of power suggesting that sUA may play an important role in self-competence and is thought to contribute to motivation and productivity. Concentration of sUA was measured from saliva collected at one time time point (arrival) prior to intervention session 1. Interpretation of values requires consideration of the context and was collected at Week 1 for exploratory comparison to other variables
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Psychosocial Treatment as Usual | Animal Assisted Intervention
Number analyzed (Participants) | 19 | 20
mg/dL | 2.80 (1.16) | 2.35 (.77)

22. Secondary Outcome: Salivary Uric Acid Level (In-session Week 4)
Description: Salivary Uric Acid (sUA) is a biomarker that may be associated with increases in blood pressure in response to stress and self-perception of power suggesting that sUA may play an important role in self-competence and is thought to contribute to motivation and productivity. Concentration of sUA was measured from saliva collected at one time time point (arrival) prior to intervention session 1. Interpretation of values requires consideration of the context and was collected at Week 4 for exploratory comparison to other variables
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Psychosocial Treatment as Usual | Animal Assisted Intervention
Number analyzed (Participants) | 19 | 20
mg/dL | 2.70 (1.18) | 2.35 (.821)

23. Secondary Outcome: Salivary Uric Acid Level (In-session Week 8)
Description: Salivary Uric Acid (sUA) is a biomarker that may be associated with increases in blood pressure in response to stress and self-perception of power suggesting that sUA may play an important role in self-competence and is thought to contribute to motivation and productivity. Concentration of sUA was measured from saliva collected at one time time point (arrival) prior to intervention session 1. Interpretation of values requires consideration of the context and was collected at Week 8 for exploratory comparison to other variables
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Psychosocial Treatment as Usual | Animal Assisted Intervention
Number analyzed (Participants) | 18 | 18
mg/dL | 2.98 (1.12) | 2.21 (.83)

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events over the course of their participation in the study (8 weeks of intervention and 8 weeks of follow up).
Arm/Group | Animal Assisted Intervention | Psychosocial Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/44/NCT05102344/Prot_SAP_001.pdf
  • Informed Consent Form (2021-08-27): https://cdn.clinicaltrials.gov/large-docs/44/NCT05102344/ICF_000.pdf